CLINICAL TRIAL: NCT07034534
Title: Effectiveness of Three Typical Yoga Poses and Conventional Physiotherapy for Kinesio Phobia Among Amateur Football Players With Chronic Ankle Instability
Brief Title: Yoga vs Deep Breathing for Kinesiophobia in Footballers With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saveetha University (Other)
Responsible Party: Principal Investigator, Snekha V, Primary investigator, Saveetha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 30/32/2024/ISRB/SR/SCPT
Record Dates: First submitted 2025-05-17; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Kinesiophobia; Chronic Ankle Instability
Keywords: Chronic ankle instability; Kinesio phobia; Mind body practice; Yoga poses; Deep breathing technique; Conventional physiotherapy; Physical and emotional stability
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three typical yoga poses and conventional physiotherapy (Active Comparator): Participants received three typical yoga poses and conventional physiotherapy for five days each, for a total of six weeks with rest periods.
  Interventions: Behavioral: Three typical yoga poses; Behavioral: Deep breathing technique
- Deep Breathing technique and conventional physiotherapy (Active Comparator): Participants received Deep Breathing technique and conventional physiotherapy for five days each, for a total of six weeks with rest periods..
  Interventions: Behavioral: Three typical yoga poses; Behavioral: Deep breathing technique

INTERVENTIONS:
Behavioral: Three typical yoga poses — duration for both group includes 10 mins 5 sec, rest period will be included
  Other Names: conventional physiotherapy
Behavioral: Deep breathing technique — duration for both group includes 10 mins 5 sec, rest period will be included
  Other Names: conventional physiotherapy

SUMMARY:
The study aimed to determine if yoga poses and conventional physiotherapy were more effective than deep breathing exercises and conventional physiotherapy in reducing kinesiophobia in amateur football players with chronic ankle instability. 28 participants were divided into an experimental and control group, with the experimental group receiving yoga poses and conventional physiotherapy, and the control group receiving deep breathing exercises and conventional physiotherapy.

DETAILED DESCRIPTION:
Yoga is an Indian mind-body practice that has become well-known all over the world. During standing, sitting, and lying supine or prone, participants' bodily motions are gradual and have a wide range of motion. It has been demonstrated that yoga practice improves balance, coordination, emotional and mental well-being which assist in increasing joint flexibility, range of motion (ROM) and muscle strength.

Three yoga poses namely, the crescent lunge pose (Halasana), warrior II pose (Virabhadrasana II), and triangle pose (Trikonasana). These yoga manoeuvres reduce pain, which enhances people's quality of life. Reports indicate that yoga alters the perception of pain and influences brain waves. Since yoga promotes both pain treatment and psychosocial healing, it has been a popular alternative pain management technique in recent years for Kinesio phobia.

Injured athletes can benefit from deep breathing as a non-pharmacological pain management technique that increases localized tissue circulation and diverts attention from their discomfort. Inducing a shift in sympathetic nervous system activity by reducing stress hormone levels and activating the diaphragm by stimulating the vagal nerve, which regulates pain perception, guided or focused deep breathing functions as a mindful meditation technique.

The most successful strategy for collegiate athletes to handle stress and prepare for competition was deep breathing. Additionally, it has been demonstrated that deep breathing can assist individuals with chronic musculoskeletal pain manage their condition effectively, reducing movement fear and enhancing subjective wellbeing and quality of life.

Conventional physical therapy includes exercises for strengthening and flexibility as well as training for agility and balance. These therapies aim to improve muscular strength, speed, agility, and neuromuscular control; restore a normal gait pattern without the use of assistive devices; improve balance; and increase range of motion and flexibility. Conventional physiotherapy uses a range of techniques centered on function restoration, strength enhancement, and injury prevention to address these problems.

By combining conventional physiotherapy with relaxation techniques like three typical yoga postures and deep breathing technique, our method not only helps people with Kinesio phobia but also improves their ankle range of motion, balance, and coordination so they can actively resume their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 22
* Acute ankle sprain diagnosis: documented diagnosis of chronic ankle instability.
* Chronic ankle instability pain score of 0-27 on CAIT tool
* Kinesio phobia severity score: 37-68 on Tampa scale
* Pain anxiety symptom scale (PASS) score: 67-94

Exclusion Criteria:

* Neurological problem
* Recent history of ankle surgery
* Proscribed with any pain - relieving medication
* Both ankle instability and acute injuries to musculoskeletal structures in the lower limb.
* Participants who have multiple fractures

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Cumberland ankle instability tool (CAIT) | Baseline and week 6
  Cumberland ankle instability tool (CAIT) is a 9-item and 30 points; self-report measures the severity of functional ankle instability. Each item has responses scored with different point values (ranging typically from 0 to 3 or 0 to 5). Total score is 30. The score from 27 to 30 represent normal stability, and the scores less than 27 representing ankle instability.
Tampa scale for kinesiophobia | Baseline and week 6
  Tampa scale is a 17-item self-reported instrument used to distinguish between non-excessive fear and phobia in patients with chronic musculoskeletal pain, i.e., the fear of movement. Each item is a 4 -point scale anchored from 1 (strongly disagree) to 4 (strongly agree) with total score of 68. The Score 17 and below representing (no kinesiophobia) and for a participants from score 37- 68 (represents kinesiophobia).

SECONDARY OUTCOMES:
Pain anxiety symptom scale | Baseline and week 6
  Pain and anxiety symptom scale (PASS) is a 20-item self-report measure to assess pain-related anxiety. Each item is a 6-point scale anchored from 0 (never) to 5 (always). Total score is ranged from 0 (representing no pain anxiety) to 100 (representing severe pain anxiety.
Y-balance test | Baseline and week 6
  The Y Balance Test (YBT) is used to assess functional equilibrium, control of posture, and lower extremity strength. In both clinical and athletic settings, it is frequently employed to evaluate injury risk, especially in patients with chronic ankle instability (CAI).

CONTACTS AND LOCATIONS:
Locations (1):
- Saveetha Institute of Medical and Technical Sciences, Chennai, Tamil Nadu, India

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT07034534/Prot_SAP_000.pdf